CLINICAL TRIAL: NCT01112449
Title: Influence of Selenium on Prostate Cancer Related Biomarkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Karam El-Bayoumy, Professor of Biochemical and Molecular Biology, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: PSHCI 08-012
Record Dates: First submitted 2010-04-23; First posted 2010-04-28 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2014-10

CONDITIONS: Effect of Selenium on Oxidative Stress in Healthy Men
Keywords: selenium; oxidative stress; prostate cancer; PSA; glucose
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Selenomethionine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Low dose selenized-yeast (Experimental): 200 µg/day of selenized-yeast (SY)
  Interventions: Dietary Supplement: low dose selenized-yeast
- selenomethionine (Experimental): The second group will receive 200 µg/day of selenomethionine (SM)
  Interventions: Dietary Supplement: selenomethionine
- Placebo (Placebo Comparator): no active medication.
  Interventions: Other: Placebo
- High dose selenized-yeast (Experimental): The fourth group will receive 285 µg/day of selenized-yeast (SY).
  Interventions: Dietary Supplement: high dose selenized-yeast

INTERVENTIONS:
Other: Placebo — no active medication
  Arms: Placebo
Dietary Supplement: selenomethionine — 200 µg/day of selenomethionine (SM)
  Other Names: SM
  Arms: selenomethionine
Dietary Supplement: low dose selenized-yeast — 200 µg/day of SY
  Other Names: low dose selenium-enriched yeast; SY
  Arms: Low dose selenized-yeast
Dietary Supplement: high dose selenized-yeast — 285 µg/day of SY
  Other Names: high dose selenium-enriched yeast; SY
  Arms: High dose selenized-yeast

SUMMARY:
Penn State Milton S. Hershey Medical Center researchers are trying to compare the effects of two different forms of selenium (selenium yeast and selenomethionine) on blood selenium levels and biomarkers of oxidative stress as primary endpoints. One in six men are at risk of getting prostate cancer in their lifetime. Participants will be asked to take over-the-counter selenium yeast supplements and selenomethionine or a placebo for nine out of twelve months.

DETAILED DESCRIPTION:
We will conduct a double-blind, randomized, placebo-controlled clinical study of selenium supplementation in the form of L-selenomethionine (SM)(200 µg/day) and selenium-enriched yeast (SY) (200 µg/day and 285 µg/day) for 9 months; the 285 µg/day SY is selected to deliver an equivalent selenium as in 200 µg/day SM to healthy men. The variability of SM in SY that will be used here is less than 3% and it accounts for 70.5% of the SM content in SY. As primary endpoints, we will determine the effects of these two forms of selenium on plasma levels of selenium and its metabolites as well as biomarkers of oxidative stress at several time points. As a secondary endpoint, the effect of these two forms of selenium on plasma PSA levels will be examined.

ELIGIBILITY:
Inclusion Criteria:

* No history or evidence of diabetes
* Male between the ages of 20-79
* PSA levels ≤ 4.0 ng/mL
* Not taking >50 µg/day selenium as a dietary supplement including multi- vitamins
* Non-smoker
* No concurrently participating or have participated in any other clinical trial within at least 30 days of registration
* Health male

Exclusion Criteria:

* Evidence of prostate cancer
* Evidence of liver or kidney disease

Ages: 20 Years to 79 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2008-05; Primary Completion 2012-07 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Biomarkers of oxidative stress | 12 months

SECONDARY OUTCOMES:
Plasma levels of selenium and selenium metabolites | 12 months
PSA | 12 months
Plasma Glucose | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Karam El-Bayoumy, PhD, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State Milton Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Derived] Richie JP Jr, Das A, Calcagnotto AM, Sinha R, Neidig W, Liao J, Lengerich EJ, Berg A, Hartman TJ, Ciccarella A, Baker A, Kaag MG, Goodin S, DiPaola RS, El-Bayoumy K. Comparative effects of two different forms of selenium on oxidative stress biomarkers in healthy men: a randomized clinical trial. Cancer Prev Res (Phila). 2014 Aug;7(8):796-804. doi: 10.1158/1940-6207.CAPR-14-0042. Epub 2014 Jun 17. PMID 24938534